CLINICAL TRIAL: NCT05333900
Title: Dietary Impact on Intestinal Sulfate Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GI-2016-25182
Record Dates: First submitted 2022-03-04; First posted 2022-04-19 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy Nutrition
Keywords: Animal-based; Plant-based; Microbiome; Hydrogen sulfide; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: 5-week crossover pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based then animal based (Active Comparator): plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Interventions: Behavioral: Plant-Based Diet then animal-based diet
- Animal-based then plant based (Active Comparator): plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Interventions: Behavioral: Animal-based diet then plant-based diet

INTERVENTIONS:
Behavioral: Plant-Based Diet then animal-based diet — Participants started with plant based diet: high in fiber, low in animal products for 7 days, with 14 day washout period between interventions. Following that, participants were switched to animal-based diet: high in animal products, low in fiber for 7 days.
  Arms: Plant-based then animal based
Behavioral: Animal-based diet then plant-based diet — Participants were started with animal-based diet: high in animal products, low in fiber for 7 days, with 14 days washout period between interventions. Following that, participants were switched to plant-based diet: high in fiber, low in animal products for 7 days
  Arms: Animal-based then plant based

SUMMARY:
This is a 5-week crossover pilot study of 15 highly motivated healthy volunteers who will consume two 7-day intervention diets: 1) a diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources; and 2) a diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources. A 14-day washout period will follow each intervention, in which participants will eat their typical diets.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Ambulatory and community dwelling
* Able and willing to comply with the study schedule and procedures
* 18 - 80 years of age
* BMI between 18.5 - 40.0 kg/m2
* Omnivorous or willing to consume animal products through duration of study

Exclusion Criteria:

* Antibiotic use within 3 months
* Planned antibiotic therapy within the period of the study, e.g., perioperative antibiotics.
* Use of sulfonamides or sulfasalazine, as these sulfur-containing medications may confound results
* Use of 5-aminosalicylates (5-ASA), as they are known to inhibit sulfidogenesis
* History of anaphylactic food allergies, e.g., peanuts, seafood.
* Food intolerances and allergies, including gluten sensitivity, lactose intolerance, and intolerance of high fiber dietary content.
* Strict vegan eating practices, with refusal to consume animal products.
* Planned use of oral probiotics while on study.
* Serious, concomitant illness that, in the opinion of the Investigator, would interfere with evaluation of safety or efficacy, or put the participant at risk of harm from study participation.
* Significant alcohol use, defined as > 20 g/day in females and > 30 g/day in males for a period of 3 months within one year prior to screening.
* Underlying chronic gastrointestinal disease that can cause diarrhea, including short bowel syndrome, irritable bowel syndrome, malabsorption, and celiac disease.
* History of partial or complete colectomy.
* History of malabsorptive bariatric surgery.
* Currently participating in another clinical study.
* Legally incompetent and unable to understand the study's purpose, significance and consequences, and to make decisions accordingly.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khoruts, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Plant-based Then Animal Based: plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources.
  animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Participants started with plant based diet: high in fiber, low in animal products for 7 days, with 14 day washout period between interventions. Following that, participants were switched to animal-based diet: high in animal products, low in fiber for 7 days.
- Animal-based Then Plant Based: plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources.
  animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Participants were started with animal-based diet: high in animal products, low in fiber for 7 days, with 14 days washout period between interventions. Following that, participants were switched to plant-based diet: high in fiber, low in animal products for 7 days
Period: Overall Study
Arm/Group | Plant-based Then Animal Based | Animal-based Then Plant Based
Started | 7 | 8
Completed | 6 | 5
Not Completed | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — COVID-19 Pandemic | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Plant-based Then Animal Based: plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Participants started with plant based diet: high in fiber, low in animal products for 7 days, with 14 day washout period between interventions. Following that, participants were switched to animal-based diet: high in animal products, low in fiber for 7 days.
- Animal-based Then Plant Based: plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
  Participants were started with animal-based diet: high in animal products, low in fiber for 7 days, with 14 days washout period between interventions. Following that, participants were switched to plant-based diet: high in fiber, low in animal products for 7 days
- Total: Total of all reporting groups
Arm/Group | Plant-based Then Animal Based | Animal-based Then Plant Based | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Effect of Short-term (1-week) Plant- and Animal-based Eating Patterns on Hydrogen Sulfide Production
Description: Determine the effect of short-term (1-week) plant- and animal-based eating patterns on ex vivo fecal hydrogen sulfide production in healthy human volunteers We will measure fecal hydrogen sulfide production ex vivo in ppm/g of dry weight of stool
Time Frame: Following 1-week of plant- and animal-based eating patterns
Measure: Median (Full Range); unit: ppm hydrogen sulfide gas
Groups:
- Plant-based Diet: plant based: diet low in sulfur-containing amino acids (Low-S diet), emphasizing plant-based foods and fat sources
- Animal-based Diet: animal based: A diet high in sulfur-containing amino acids (High-S diet), emphasizing animal protein and fat sources
Arm/Group | Plant-based Diet | Animal-based Diet
Number analyzed (Participants) | 11 | 11
ppm hydrogen sulfide gas | 69 [7.5 to 217.5] | 103 [27.7 to 286.9]

ADVERSE EVENTS:
Time Frame: 6-weeks
Arm/Group | Plant-based Diet | Animal-based Diet
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT05333900/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT05333900/ICF_001.pdf